CLINICAL TRIAL: NCT06133413
Title: Connected Scales to Optimize the Maintenance of Weight Lost After Bariatric Surgery and Limit Failures and Reoperations
Acronym: COMPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Withings (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP230777
Record Dates: First submitted 2023-10-30; First posted 2023-11-15 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Obesity, Severe; Surgery
Keywords: Obesity surgery; Connected scale; Remote patient monitoring
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: Comparative, controlled, randomized 1:1, open, in two parallel arms study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care group (No Intervention): Standard follow-up
- Connected scale group (Experimental): Standard follow up + Use weekly of Body Comp Pro connected scale, associated with a remote monitoring by medical team allowing alert generation and early intervention
  Interventions: Device: Body Comp Pro connected scale (Withings manufacturer); Other: Alert generation by remote plateform

INTERVENTIONS:
Device: Body Comp Pro connected scale (Withings manufacturer) — Use once a week
  Arms: Connected scale group
Other: Alert generation by remote plateform — Alert will be generated from weight regain > 5% of baseline weight
  Arms: Connected scale group

SUMMARY:
In this research, we hypothesize that post-operative monitoring implemented with a connected scale after the 1st year (weight nadir period) post obesity surgery (i.e. sleeve and RYGB) would reduce the percentage of patients with excessive weight regain (>10% regain of lost weight) by improving the quality of follow-up and long-term results.

To do this, we are carrying out a comparative study on 182 patients, controlled, randomized per patient, ratio 1/1, open, in two parallel arms.

Patients will be followed for 12 months and divided into one of the following two groups:

* Control group: Standard follow-up
* Interventional group: Standard follow-up + weekly weighing with the "Body Comp Pro" connected scale

During their follow-up period, patients in the intervention group will have to weigh themselves at least once a week using the "Body Comp Pro" connected scale. The information will be transmitted to the investigation team via a secure platform available 24 hours a day. Alerts will be generated from a weight regain > 5% of the baseline weight, allowing early management of weight regain.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged 18 and over
* Patient operated by a sleeve or RYGB at 1 year (+/- 1 month) from the inclusion visit
* Patient affiliated to a social security system (excluding AME)
* Patient having signed free, informed and written consent
* Patient speaking and reading French fluently

Exclusion Criteria:

* Patient with medical-surgical complications during inclusion visit justifying specific and reinforced monitoring (at the discretion of the investigator)
* Patient with a pacemaker
* Patient with a pathology or disability preventing them from standing on the scale
* Patient participating in another interventional research at the time of inclusion
* At the interview, pregnant patient or planning pregnancy during her period of participation in the research
* Patient deprived of liberty
* Patient subject to a legal protection measure (guardianship, curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Compare the percentage of patients with weight regain > 10% at 24 months post-operative in patients who have undergone obesity surgery (SG or RYGB) in the two groups of patients | 12 months from inclusion
  Percentage of patients with weight regain > 10% between inclusion (12 months post-op) and the 12-month visit (24 months post-op) in the two groups of patients

SECONDARY OUTCOMES:
To compare the weight change at 18 and 24 months post-operative in patients having undergone obesity surgery (SG or RYGB) in the two groups of patients | 6 and 12 months from inclusion
  Weight change (in kilos and % of weight lost since the intervention) between the weight at inclusion (12 months post-op) and the weight at 6 and 12 months from inclusion (18 and 24 months post-op ) in both groups of patients.
To compare the number of surgical reinterventions (planned or carried out) for weight regain at 24 months post-operative in patients having undergone obesity surgery (SG or RYGB) in the two groups of patients | 12 months from inclusion
  Number of surgical reinterventions (planned or carried out) for excessive weight gain validated in a multidisciplinary consultation meeting between inclusion (12 months post-op) and the visit 12 months from inclusion (24 months post-op) in both patient groups
To compare the evolution of comorbidities at 18 and 24 months post-operative in patients having undergone obesity surgery (SG or RYGB) in the two groups of patients | 6 and 12 months from inclusion
  Resolution, evolution, recurrence, or occurrence of a comorbidity between inclusion (12 months post-op) and visits at 6 and 12 months from inclusion (18 and 24 months post-op) in the two groups of patients. The comorbidities identified are High blood pressure, Type 2 diabetes and sleep apnea syndrome
To compare anxiety and depression at 18 and 24 months post-operative in patients having undergone obesity surgery (SG or RYGB) in the two groups of patients | 6 and 12 months from inclusion
  Evolution of the HAD scale score between inclusion (12 months post-op) and visits at 6 and 12 months from inclusion (18 and 24 months post-op) in the two groups of patients
Compare the quality of life at 18 and 24 months post-operative in patients having undergone obesity surgery (SG or RYGB) in the two groups of patients | 6 and 12 months from inclusion
  Evolution of the SF-36 quality of life score between inclusion (12 months post-op) and visits at 6 and 12 months from inclusion (18 and 24 months post-op) in the two groups of patients
Compare the number of lost to follow-up at 18 and 24 months post-operative in patients having undergone obesity surgery (SG or RYGB) in the two groups of patients | 6 and 12 months from inclusion
  Number of patients lost to follow-up between inclusion (12 months post-op) and visits at 6 and 12 months from inclusion (18 and 24 months post-op) in the two groups of patients
To compare the change in body composition measured by a connected scale at 18 and 24 months post-operative in patients having undergone obesity surgery (SG or RYGB) in the two groups of patients | 6 and 12 months from inclusion
  Evolution of body composition (muscle mass, fat mass) measured by the connected scale between the inclusion visit (12 months post-op) and the visits at 6 and 12 months from inclusion (18 and 24 months post-op ) in both groups of patients.
For interventionnal group only : Evaluate the impact of the use of a connected scale on the consumption of additional care at 18 and 24 months post-operative in patients having undergone obesity surgery (SG or RYGB). | 6 and 12 months from inclusion
  Number of telephone calls, consultations or hospitalizations in hospital, secondary to an alert generated by the connected scale between the inclusion visit (12 months post-op) and the visits at 6 and 12 months of inclusion (18 and 24 months post-op) for each patient in the interventional group
For interventionnal group only : Evaluate adherence to the use of a connected scale at 18 and 24 months post-operative in patients having undergone obesity surgery (SG or RYGB) | 6 and 12 months from inclusion
  Average frequency of use of the connected scale between inclusion (12 months post-op) and visits at 6 and 12 months from inclusion (18 and 24 months post-op) for each patient in the interventional group compared to this which is required of them (i.e. 1 weighing per week)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital La Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No